CLINICAL TRIAL: NCT03944226
Title: Is Dietary Nitrate Effective in Reducing Aerobic Glycolysis (AG) in Breast Cancer? - A Longitudinal Study Using Specialist Magnetic Resonance (MR) Methods
Brief Title: Is Dietary Nitrate Effective in Reducing Aerobic Glycolysis in Breast Cancer?
Acronym: BEET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2-114-18; 17/049 (Other Grant/Funding Number: Research and Development Endowment Research Grants)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Malignant Breast Tissue Neoplasm
Keywords: Beetroot juice; Magnetic Resonance Imaging; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group: trials with a single arm
Masking Description: Single group with no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beetroot (Experimental): 16 patients confirmed with a diagnosis of invasive ductal carcinoma who will undergo wide local excision surgery or mastectomy. All patients in the single arm will undergo a 5 day intervention drinking concentrated beetroot juice and 2 magnetic resonance imaging scan sessions pre and post intervention. MRI scan sessions will be composed of research scans including diffusion and lipid profiling MR imaging methods and MR spectroscopy (MRS) methods.
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — The patient will follow a 5 day dietary nitrate intervention programme, taking 3 doses of 7cl (0.4 g nitrate per dose) concentrated beetroot juice (SPORT shot, James White Drinks, Suffolk, U.K.) a day.

SUMMARY:
Breast cancer is the most prevalent cancer affecting women, with 1 in 8 women in the UK developing breast cancer in their life time. Chemotherapy drugs, currently used for locally advanced breast cancers, are associated with side effects while dietary supplements have complex effects with a relatively small effect size.

Breast tumours have different metabolism compared to healthy tissue, including elevated lactate production by aerobic glycolysis (AG), an underpinning feature of metabolism in breast cancer cells. Dietary nitrate, contained in leafy green vegetables and beetroot, has been shown to improve energy efficiency in exercising skeletal muscle, positioning itself as a disruptor of AG.

The purpose of this study is to examine if dietary nitrate can disrupt AG and as a result to halt or even reverse tumour progression and survival. This study will look at scans of breast tumours using magnetic resonance imaging (MRI). Changes to tumour related biochemical substances will be measured by advanced magnetic resonance spectroscopy and changes to tissue structure will be measured by advanced diffusion MRI techniques.

In this study, 16 patients undergoing surgery will be recruited for two MRI scans following a 5 day intervention programme.

DETAILED DESCRIPTION:
In this longitudinal study, the investigators propose to examine the changes in lipid composition and microstructure in breast tumours at baseline and post dietary nitrate intervention through the applications of novel non-invasive magnetic resonance spectroscopy (MRS) methods and diffusion and lipid profiling MR imaging methods in patients. The investigators hypothesise that dietary nitrate disrupts tumour progression in breast cancer.

1. Is there a significant difference in lipid composition in the tumour measured by MRS between baseline and post dietary nitrate intervention?
2. Is there a significant difference in lipid composition in the whole breast tissue surrounding tumour measured by MRI between baseline and post dietary nitrate intervention?
3. Is there a significant difference in tissue microstructure measured by MRI between baseline and post dietary nitrate intervention in the breast tissue?

To assess the effect of dietary nitrate on tumour progression, paired t-tests will be performed on lipid composition measured from tumour between baseline and post intervention. To assess the effect of dietary nitrate on tumour progression, paired t-tests will be performed on lipid composition in the whole breast tissue surrounding tumour between baseline and post intervention. To assess the effect of dietary nitrate on tissue microstructure paired t-tests will be performed on water displacement measured from tumour between baseline and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed invasive ductal carcinoma (Grade 2 or 3)
* Undergoing wide local excision surgery or mastectomy

Exclusion Criteria:

* Started hormone or chemotherapy treatment before recruitment.
* Undergoing treatment for concurrent cancer diagnosis.
* Taking antibiotics, proton pump or vegetable dietary supplement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-05-13 (Estimated); Primary Completion 2020-04-26 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline: Lipid composition in tumour | Scan one day before intervention (Day 0)
  Lipid peak volume with units of ratio
Post intervention: Lipid composition in tumour | Scan one day after completion of intervention (Day 6)
  Lipid peak volume ratio with units of ratio
Baseline: Lipid composition in whole breast tissue surrounding tumour | Scan one day before intervention (Day 0)
  fat fraction with units of %
Post intervention: Lipid composition in whole breast tissue surrounding tumour | Scan one day after completion of intervention (Day 6)
  fat fraction with units of %
Baseline: Water displacement in tumour | Scan one day before intervention (Day 0)
  Water displacement with units of micrometer
Post intervention: Water displacement in tumour | Scan one day after completion of intervention (Day 6)
  Water displacement with units of micrometer

CONTACTS AND LOCATIONS:
Overall Officials: Jiabao He, PhD, Study Chair — University of Aberdeen; Vasiliki Mallikourti, MSc, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Biomedical Imaging Centre, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham LJ, Shupe MP, Schneble EJ, Flynt FL, Clemenshaw MN, Kirkpatrick AD, Gallagher C, Nissan A, Henry L, Stojadinovic A, Peoples GE, Shumway NM. Current approaches and challenges in monitoring treatment responses in breast cancer. J Cancer. 2014 Jan 5;5(1):58-68. doi: 10.7150/jca.7047. PMID 24396498
- [Background] Baker J, Ajani J, Scotte F, Winther D, Martin M, Aapro MS, von Minckwitz G. Docetaxel-related side effects and their management. Eur J Oncol Nurs. 2009 Feb;13(1):49-59. doi: 10.1016/j.ejon.2008.10.003. Epub 2009 Feb 7. PMID 19201649
- [Background] Gatenby RA, Gillies RJ. Why do cancers have high aerobic glycolysis? Nat Rev Cancer. 2004 Nov;4(11):891-9. doi: 10.1038/nrc1478. PMID 15516961
- [Background] Jones AM. Dietary nitrate supplementation and exercise performance. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S35-45. doi: 10.1007/s40279-014-0149-y. PMID 24791915
- [Background] McMahon NF, Leveritt MD, Pavey TG. The Effect of Dietary Nitrate Supplementation on Endurance Exercise Performance in Healthy Adults: A Systematic Review and Meta-Analysis. Sports Med. 2017 Apr;47(4):735-756. doi: 10.1007/s40279-016-0617-7. PMID 27600147
- [Background] Bentley R, Gray SR, Schwarzbauer C, Dawson D, Frenneaux M, He J. Dietary nitrate reduces skeletal muscle oxygenation response to physical exercise: a quantitative muscle functional MRI study. Physiol Rep. 2014 Jul 22;2(7):e12089. doi: 10.14814/phy2.12089. Print 2014 Jul 1. PMID 25052493